CLINICAL TRIAL: NCT05018988
Title: The D-VinCHI Study: 25-hydroxyvitamin D Concentration in School Children: Effects of Vitamin D3 Supplementation on 25-OH-D Concentration and Muscle Health Outcomes
Brief Title: Vitamin D in School Children
Acronym: DVinCHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Queen Margaret University, Nutrition and Biological Sciences, Musselburgh, Scotland, UK (Unknown); Better You ltd., Unit 24 Shortwood Court, Shortwood Business Park, Dearne Valley Parkway, Barnsley, S74 9LH, Registered Company No: 05541287 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DVinCHI_UU2019
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D Deficiency; Musculoskeletal Diseases; Cognitive Delay, Mild
Keywords: Vitamin D; Deficiency; vitamin D3; supplementation; Cholecalciferol; school children; paediatric; 25(OH)D; hypovitaminosis D; postural balance; cognitive function
MeSH Terms: conditions — Vitamin D Deficiency; Musculoskeletal Diseases; Lymphoma, Follicular | interventions — Cholecalciferol; Xylitol

STUDY DESIGN:
Intervention Model Description: Observational study followed double blinded randomised control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded to participant and researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral vitamin D3 spray (Experimental): 10µg/day for 12 weeks (BetterYou ltd.)
  Interventions: Dietary Supplement: Oral vitamin D spray
- Placebo Comparator (Placebo Comparator): Xylitol (BetterYou ltd.)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral vitamin D spray — 1 spray (10µg) /day for 12 weeks
  Other Names: vitamin D3
  Arms: Oral vitamin D3 spray
Dietary Supplement: Placebo — 1 spray / day for 12 weeks
  Other Names: Xylitol
  Arms: Placebo Comparator

SUMMARY:
The primary purpose of this study it to investigate total circulating 25-hydroxyvitamin D (25(OH)D) in school children (aged 4-11years) in Northern Ireland; thereby establishing the prevalence of vitamin D status (deficiency, insufficiency, and sufficiency (SACN 2016)) in this cohort. Additionally, the study aims to determine if 10µg/day vitamin D3 supplementation over 12 weeks maintains vitamin D status.

This area of research is lacking in the quality of prospective studies. While previous literature has focused on the prevalence of vitamin D status in adults, there is a paucity of data available for children. This study will add to the existing knowledge and provide more specific analysis for children.

Hypothesis 1: Increase in vitamin D concentrations will be associated with an improvement in health outcomes including anthropometric measurements, musculoskeletal outcomes, markers of inflammation, nutritional status and bone turnover, lipid profiles, cognitive function, and handgrip strength.

DETAILED DESCRIPTION:
The main objectives of this study are to determine prevalence of vitamin D status in 4-11-year-old children and to investigate if 10µg/day maintains vitamin D status in this population. This study will focus on children aged 4-11 years old residing in Northern Ireland. This 2-phase study will incorporate an observational phase and intervention phase to determine prevalence and status, respectively. The expected time under study will be 12 weeks and the number of visits will be limited to two per participant. Where participants are from the same home, randomisation to the same treatment group will occur. Results will be controlled for season.

Vitamin D deficiency is prevalent across the global population including those who reside above 37° North. In addition to a lack of rich dietary sources of vitamin D, residing at this latitude restricts exposure to sunlight due to the zenith angle of the sun. Although vitamin D deficiency is rife in the general population there are certain categories who are at additional risk of vitamin D deficiency including pregnant women, elderly, and institutionalized populations. One population group where there is still a paucity of studies, and a lack of clear guidelines are children. Recent evidence suggests that vitamin D has potential to provide extra skeletal health benefits.

Assessments to be undertaken in this study include anthropometric, handgrip, balance, cognitive function. These assessments will be followed by a 20ml blood draw completed by a trained researcher who is trained in phlebotomy. Additionally, parents will be asked to complete a validated vitamin D food frequency questionnaire and four-day weighed diet diary for their offspring. This study will determine if the recommended supplementation regimen results in the intervention population reporting a sufficient vitamin D status. Blood samples will be analysed for 25(OH)D, serum parathyroid hormone (PTH), serum C-reactive protein (CRP), serum HbA1c (glycated haemoglobin), markers of bone turnover, markers of inflammation, full blood count, lipid profile, and markers of nutritional status. Circulating 25(OH)D will be assessed via liquid chromatography- mass spectrometry (HPLC & MS).

Sample size was calculated using G*Power software available at QMU (G*Power) by entering the planned statistical analysis method (i.e. t-test or ANOVA), desired effect size (0.5), and experimental design (i.e. two groups with two outcomes). Phase one (observational study) with an effect size of 0.15 requires a total population of 200. Phase two (intervention study) with an effect size of 0.15 requires a total population of 118 (59 in each arm) including a dropout rate of 20%. A total population of 55 is required for Food frequency validation including a 10% dropout rate and for the vitamin D knowledge questionnaire with an effect size of 0.8 a total population of 70 is required.

The planned statistical analysis will be conducted in IBM SPSS and with intention to treat. Results from phase one will be analysed using descriptive statistics. A regression model will be used to determine prediction models for circulating 25(OH)D and the reported secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 4-11 years attending school in Northern Ireland.

Exclusion Criteria:

* Any children on long-term prescription medication; and/or diagnosed with a long-term or exacerbated health condition or disease (does not exclude children with minor or mild health conditions).
* Those previously taking a vitamin D supplement and those not willing to abstain from starting vitamin D supplements.
* Those using home sun beds.
* Those who are planning a family holiday to a sunny country (latitudes below 37°N) during the duration of the intervention.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Plasma 25-hydroxy vitamin D concentration | Change over 12 weeks
  Measured by LC/MS

SECONDARY OUTCOMES:
Muscle strength | Change over 12 weeks
  Hand grip strength by a dynamometer
Postural balance | Change over 12 weeks
  Assessed using single leg stance (SLS)
Postural balance | Change over 12 weeks
  Assessed using tandem stance (TS)
Cognitive function | Change over 12 weeks
  Assessed using three CANTAB batteries

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Londonderry, United Kingdom